CLINICAL TRIAL: NCT00287196
Title: Randomised Clinical Trial of Surgery Versus Surgery Plus Adjuvant Radiotherapy for Regional Control in Patients With Completely Resected Macroscopic Nodal Metastatic Melanoma
Brief Title: Immediate Radiotherapy or Observation After Surgery for Melanoma Involving Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: University Medical Center Groningen (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 02.01; NHMRC 251732 (Other Grant/Funding Number: NHMRC); ANZMTG 01.02 (Other: Austalian NewZealand Melanoma Trials Group)
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2009-09

CONDITIONS: Malignant Melanoma; Lymph Node Disease
Keywords: Melanoma; Lymph node disease; Adjuvant radiotherapy; Lymphoedema
MeSH Terms: conditions — Melanoma; Lymphedema | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-operative RADIOTHERAPY (Active Comparator): Immediate post-operative RADIOTHERAPY
  Interventions: Radiation: Radiotherapy
- Delayed Radiotherapy (Experimental): OBSERVATION with delayed radiotherapy for relapse
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 48 Gy reference dose in 20 fractions at 5 fractions per week, with a maximum overall treatment time of 30 days.
  Other Names: Radiation

SUMMARY:
This trial seeks to establish the role of post-operative radiotherapy in patients who have had surgery for melanoma involving lymph nodes and who are at high risk of recurrence.

DETAILED DESCRIPTION:
This is a randomised phase III trial which is being performed on patients at high risk of local recurrence after having a lymphadenectomy for stage 3 melanoma. The control arm is surgery alone with radiotherapy reserved for those who recur. The study arm is surgery plus post-operative radiotherapy. All 3 major node sites are eligible. The radiation dose administered is 48Gy in 20 fractions. It is likely to be the only study of its kind ever performed. The target is 230 patients.

ELIGIBILITY:
Inclusion Criteria:

* Regional macroscopic nodal metastatic melanoma in one nodal basin region only which has been completely resected.
* melanoma involving lymph nodes at high risk of local recurrence (details in protocol)
* No evidence of metastases
* No active major cancer within 5 years
* Normal blood tests
* WHO performance status of 0 or 1
* Radiotherapy must be able to be commenced within 12 weeks of lymphadenectomy
* Patient must not be pregnant and if fertile must use a medically acceptable contraceptive throughout treatment
* No major concurrent illnesses likely to cause death within 2 years
* Written informed consent has been given

Exclusion Criteria:

* Evidence of active or previous local recurrence or in transit disease
* Evidence of distant metastases on clinical or radiological investigation
* Patients with prior cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2002-03; Primary Completion 2008-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Locoregional control | Final analysis will occur when all patients have had 1 year follow up. (approx. 7 years after start of trial)

SECONDARY OUTCOMES:
Disease-free survival | Final analysis will occur when all patients have had 1 year follow up. (approx. 7 years after start of trial)
Overall survival | Final analysis will occur when all patients have had 1 year follow up. (approx. 7 years after start of trial)
Toxicity | Interim analysis will occur on annual basis.
Quality of life | Final analysis will occur when all patients have had 1 year follow up. (approx. 7 years after start of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Burmeister, Study Chair — Princess Alexandra Hospital
Locations (22):
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Mater Hospital - North sydney, Crows Nest, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Hospital do Cancer, São Paulo, Brazil
- Groningen University Hospital, Groningen, Netherlands
- New Zealand (4):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Wellington

REFERENCES:
- [Derived] Henderson MA, Burmeister BH, Ainslie J, Fisher R, Di Iulio J, Smithers BM, Hong A, Shannon K, Scolyer RA, Carruthers S, Coventry BJ, Babington S, Duprat J, Hoekstra HJ, Thompson JF. Adjuvant lymph-node field radiotherapy versus observation only in patients with melanoma at high risk of further lymph-node field relapse after lymphadenectomy (ANZMTG 01.02/TROG 02.01): 6-year follow-up of a phase 3, randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1049-1060. doi: 10.1016/S1470-2045(15)00187-4. Epub 2015 Jul 20. PMID 26206146
- [Derived] Burmeister BH, Henderson MA, Ainslie J, Fisher R, Di Iulio J, Smithers BM, Hong A, Shannon K, Scolyer RA, Carruthers S, Coventry BJ, Babington S, Duprat J, Hoekstra HJ, Thompson JF. Adjuvant radiotherapy versus observation alone for patients at risk of lymph-node field relapse after therapeutic lymphadenectomy for melanoma: a randomised trial. Lancet Oncol. 2012 Jun;13(6):589-97. doi: 10.1016/S1470-2045(12)70138-9. Epub 2012 May 9. PMID 22575589
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au